CLINICAL TRIAL: NCT01256294
Title: A Prospective, Multi-center, Open-label, Randomized, Two Period, Two Sequence, Crossover Study to Compare the Steady State Pharmacokinetics of Generic Tacrolimus (Sandoz) to Prograf in Stable Renal Transplant Patients
Brief Title: Pharmacokinetics of Generic to Brand Tacrolimus in Stable Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AUS90
Record Dates: First submitted 2010-11-01; First posted 2010-12-08 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-05

CONDITIONS: Renal Transplant
Keywords: Renal transplant; kidney transplant; immunosuppressive therapy; anti-rejection medication; pharmacokinetics; tacrolimus
MeSH Terms: interventions — Tacrolimus

ARMS (2):
- Sequence 1 - Branded Tacrolimus / Generic Tacrolimus (Experimental): In Period 1 (Days 1-14) participants received branded tacrolimus (Prograf) orally twice a day and in Period 2 (Days 15 - 28) participants received generic tacrolimus (Sandoz) orally twice a day. Participants received the same stable dosage of tacrolimus they had been taking prior to enrollment (on a milligram for milligram basis).
  Interventions: Drug: Generic Tacrolimus; Drug: Branded Tacrolimus
- Sequence 2 - Generic Tacrolimus / Branded Tacrolimus (Active Comparator): In Period 1 (Days 1 - 14) participants received generic tacrolimus (Sandoz) orally twice a day and in Period 2 (Days 15 - 28) participants received branded tacrolimus (Prograf) orally twice a day. Participants received the same stable dosage of tacrolimus they had been taking prior to enrollment (on a milligram for milligram basis).
  Interventions: Drug: Generic Tacrolimus; Drug: Branded Tacrolimus

INTERVENTIONS:
Drug: Generic Tacrolimus — Generic Sandoz tacrolimus supplied as capsules of 0.5 mg, 1 mg and 5 mg dose strengths.
  Other Names: Sandoz
Drug: Branded Tacrolimus — Capsules supplied at dose strengths of 0.5 mg, 1 mg, and 5 mg.
  Other Names: Prograf

SUMMARY:
The study is designed to compare the pharmacokinetics of generic tacrolimus (Sandoz) to branded tacrolimus (Prograf) in stable renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate and willing to give written informed consent and to comply with the study visits and restrictions.
* Patient who has received a primary or secondary kidney transplant
* Patient who is at least 6 months post transplant and on a stable dose of tacrolimus as defined by physician, one tacrolimus trough level within the physician defined target range within past 6 months and one additional trough level during the screening period within 30% of the physician defined target range.
* Body mass index (BMI) greater than or equal to 19 but less than or equal to 35
* Patients who are taking tacrolimus (generic, Sandoz) or Prograf

Exclusion Criteria:

* Evidence of any acute rejection
* Patients who require dialysis within 6 months prior to study entry
* Recipients of antibodies blood group (ABO) incompatible allograft or positive crossmatch
* Recipients of multiple organ transplants
* Patients who have tested positive for hepatitis B surface antigen (HBsAG) or human immunodeficiency virus (HIV), or who are recipients of organ from donors who are known to be HBsAG or HIV positive. Virology screening at the time of transplant was acceptable unless more recent tests were available.
* History of malignancy, treated or untreated, within the past 2 years with the exception of carcinoma in situ or excised basal cell carcinoma
* Glomerular filtration rate ≤35 ml/min measured by modification of diet in renal disease (MDRD4)
* No anticipated change in the immunosuppressive regimen during patient participation other than that required by the protocol
* Initiation of any medications that could interfere with tacrolimus blood levels, including over the counter medications, herbal supplements, grapefruit or grapefruit juice.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are

  * women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner
  * women whose partners have been sterilized by vasectomy or other means
  * using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices (IUDs); periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.
* Patients who are taking a generic tacrolimus product other than tacrolimus (generic, Sandoz).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 - Branded Tacrolimus / Generic Tacrolimus: In Period 1 (Days 1 - 14) participants received branded tacrolimus (Prograf) orally twice a day and in Period 2 (Days 15 - 28) participants received generic tacrolimus (Sandoz) orally twice a day. Participants received the same stable dosage of tacrolimus they had been taking prior to enrollment (on a milligram for milligram basis).
- Sequence 2 - Generic Tacrolimus / Branded Tacrolimus: In Period 1 (Days 1-14) participants received generic tacrolimus (Sandoz) orally twice a day and in Period 2 (Days 15-28) participants received branded tacrolimus (Prograf) orally twice a day. Participants received the same stable dosage of tacrolimus dose they had been taking prior to enrollment (on a milligram for milligram basis).
Period: Overall Study
Arm/Group | Sequence 1 - Branded Tacrolimus / Generic Tacrolimus | Sequence 2 - Generic Tacrolimus / Branded Tacrolimus
Started | 36 | 35
Completed | 32 | 33
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol deviation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Period 1 (Days 1 through 14): Participants randomized to Sequence 1 took branded tacrolimus (Prograf) and participants randomized to Sequence 2 took generic tacrolimus (Sandoz).
  Period 2 (Days 15 through 28): Participants randomized to Sequence 1 crossed over to treatment with generic tacrolimus and participants randomized to Sequence 2 crossed over to treatment with branded tacrolimus.
Arm/Group | All Participants
Number analyzed (Participants) | 71
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Dose-Normalized Area Under the Concentration-time Curve From Time 0 to 12 Hours (AUC0-12h) at Steady State
Description: Dose-normalized area under the concentration-time curve from time 0 to 12 hours (AUC0-12h) at steady state after 14 days of treatment with each study drug.
  Geometric mean and 95% confidence intervals were determined from an analysis of variance (ANOVA) model for the dose-normalized log transformed values with treatment, period and sequence as fixed factors and patients nested within sequences as a random factor.
Time Frame: Days 14 and 28: Predose and at 0.5, 1, 1.5, 1.75, 2, 3, 4, 8 and 12 hours after dosing.
Population: Pharmacokinetic (PK) analysis set included the subset of patients from the Full Analysis Set (all patients to whom study medication had been assigned) with evaluable PK data.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL/mg
Groups:
- Generic Tacrolimus: Participants received generic tacrolimus (Sandoz) orally twice a day for 14 days.
- Branded Tacrolimus: Participants received branded tacrolimus (Prograf) orally twice a day for 14 days.
Arm/Group | Generic Tacrolimus | Branded Tacrolimus
Number analyzed (Participants) | 65 | 66
ng*hr/mL/mg | 51.73 [44.67 to 59.90] | 50.58 [43.68 to 58.57]
Statistical Analysis 1: Comparison: Generic Tacrolimus vs Branded Tacrolimus; Test type: Superiority or Other; Ratio of geometric means = 1.02, 95% CI 2-sided [0.96 to 1.09]
Statistical Analysis 2: Comparison: Generic Tacrolimus vs Branded Tacrolimus; To compare the bioavailability of generic tacrolimus to branded tacrolimus, the 90% confidence intervals of the ratios of geometric means of AUC0-12h were assessed relative to the interval [80%, 125%]; Test type: Superiority or Other; p = 0.486, ANOVA — ANOVA model for the dose-normalized log transformed values with treatment, period and sequence as fixed factors and subjects nested within sequences as a random factor; Ratio of geometric means = 1.02, 90% CI 2-sided [0.97 to 1.08]

2. Secondary Outcome: Intra-patient Variability of Tacrolimus Pharmacokinetic Parameters
Description: The intra-patient variability of tacrolimus pharmacokinetics of each formulation was evaluated by comparing AUC0-12h, maximum drug concentration (Cmax) and trough drug concentration (C0) at Days 7 and 14, and Days 21 and 28. Intra-patient variability was assessed by a calculation of the coefficient of variation, by patient, using the repeated measurements within each Period, where the coefficient of variation (%) = standard deviation/mean*100.
Time Frame: Days 7 and 14, and Days 21 and 28.
Population: PK Analysis set.
Measure: Mean (Standard Error); unit: percent coefficient of variation
Arm/Group | Generic Tacrolimus | Branded Tacrolimus
Number analyzed (Participants) | 65 | 66
percent coefficient of variation
  AUC0-12h | 13.41 (10.438) | 11.02 (9.756)
  Cmax | 16.92 (15.485) | 17.86 (14.874)
  C0 | 13.24 (9.766) | 11.07 (10.285)

3. Secondary Outcome: Trough Plasma Drug Concentration (C0) at Steady State
Description: Trough plasma drug concentration measured prior to drug administration at steady state (after 14 days of treatment with each study drug).
Time Frame: Days 14 and 28: predose
Population: PK analysis set, where data were available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Generic Tacrolimus | Branded Tacrolimus
Number analyzed (Participants) | 65 | 66
ng/mL
  Day 14 [N= 34, 33] | 7.25 (1.580) | 7.01 (1.694)
  Day 28 [N=31, 33] | 7.26 (2.091) | 7.04 (2.379)

4. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was defined as the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event was not considered to be related to study drug. An SAE was an event which: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; required or prolonged inpatient hospitalization; was medically significant, i.e., an event that jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: 28 Days
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Generic Tacrolimus | Branded Tacrolimus
Number analyzed (Participants) | 71 | 71
participants
  Any adverse event | 8 | 12
  Serious adverse event | 0 | 1

5. Secondary Outcome: Number of Participants With Reported Biopsy Proven Acute Rejection Episodes
Time Frame: 28 Days
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Generic Tacrolimus | Branded Tacrolimus
Number analyzed (Participants) | 71 | 71
participants | 0 | 0

6. Primary Outcome: Dose-normalized Maximum Plasma Drug Concentration (Cmax) at Steady State
Description: Maximum (peak) plasma drug concentration after drug administration at steady state (after 14 days of treatment with each study drug). Geometric mean and 95% confidence intervals were determined from an analysis of variance (ANOVA) model for the dose-normalized log transformed values with treatment, period and sequence as fixed factors and patients nested within sequences as a random factor.
Time Frame: Days 14 and 28: Predose and at 0.5, 1, 1.5, 1.75, 2, 3, 4, 8 and 12 hours after dosing.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Generic Tacrolimus | Branded Tacrolimus
Number analyzed (Participants) | 65 | 66
ng/mL/mg | 8.34 [7.24 to 9.61] | 7.62 [6.61 to 8.78]
Statistical Analysis 1: Comparison: Generic Tacrolimus vs Branded Tacrolimus; Test type: Superiority or Other; Ratio of geometric means = 1.09, 95% CI 2-sided [1.00 to 1.20] — Ratio of geometric means: Generic tacrolimus/Branded tacrolimus
Statistical Analysis 2: Comparison: Generic Tacrolimus vs Branded Tacrolimus; To compare the bioavailability of generic tacrolimus to branded tacrolimus, the 90% confidence intervals of the ratios of geometric means of Cmax were assessed relative to the interval [80%, 125%]; Test type: Superiority or Other; p = 0.057, ANOVA — [p-value comment as in outcome 1, analysis 2]; Ratio of geometric means = 1.09, 90% CI 2-sided [1.01 to 1.18]

ADVERSE EVENTS:
Arm/Group | Generic Tacrolimus | Branded Tacrolimus
Serious Adverse Events (participants affected / at risk) | 0/71 | 1/71
Other Adverse Events (participants affected / at risk) | 0/71 | 4/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Tacrolimus (N=71) | Branded Tacrolimus (N=71)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Tacrolimus (N=71) | Branded Tacrolimus (N=71)
Vomiting (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.